CLINICAL TRIAL: NCT05364047
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Immunogenicity of SARS-CoV-2 mRNA Vaccine (LVRNA009) in Chinese People Aged 18 Years and Over
Brief Title: Clinical Trial of SARS-CoV-2 mRNA Vaccine in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: Shulan (Hangzhou) Hospital (Other); Yuncheng Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LVRNA009-I-01
Record Dates: First submitted 2022-04-22; First posted 2022-05-06 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — LVRNA009 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low-dose group, 18-59 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 25μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: Low-dose of LVRNA009; Other: Placebo
- Middle-dose group, 18-59 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 50μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: Middle-dose of LVRNA009; Other: Placebo
- High-dose group, 18-59 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 100μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: High-dose of LVRNA009; Other: Placebo
- Low-dose group, over 60 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 25μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: Low-dose of LVRNA009; Other: Placebo
- Middle-dose group, over 60 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 50μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: Middle-dose of LVRNA009; Other: Placebo
- High-dose group, over 60 years of age (Other): The subjects were divided into the experimental group and the placebo group according to 3:1. The experimental group was inoculated with a dose of 100μg mRNA vaccine, and the placebo group was inoculated with a dose of placebo.
  Interventions: Biological: High-dose of LVRNA009; Other: Placebo

INTERVENTIONS:
Biological: Low-dose of LVRNA009 — 25μg/person
  Arms: Low-dose group, 18-59 years of age; Low-dose group, over 60 years of age
Biological: Middle-dose of LVRNA009 — 50μg/person
  Arms: Middle-dose group, 18-59 years of age; Middle-dose group, over 60 years of age
Biological: High-dose of LVRNA009 — 100μg/person
  Arms: High-dose group, 18-59 years of age; High-dose group, over 60 years of age
Other: Placebo — 0.5ml/person

SUMMARY:
This study is a phase I clinical trial. The investigators intent to evaluate the safety, tolerability and preliminary immunogenicity of SARS-CoV-2 mRNA vaccine (LVRNA009) in Chinese people aged 18 years and over.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of the first dose of vaccine: aged 18 to 59 years (including boundary values) in the adult group, >=60 years old in the older group, regardless of gender;
2. Axillary body temperature is less than 37.3 ℃ on the day of enrollment;
3. Based on the medical history and relevant physical examination and laboratory examination results, the investigator clinically determined that the patient was in good health;
4. Subjects have independent judgment ability, can read, understand and complete vaccination diary cards, and they participate voluntarily and sign an informed consent form.

Exclusion Criteria:

1. The subject has a history of SARS-CoV-2 infection, or has a history of contact with SARS-CoV-2 infected persons (nucleic acid test positive) or suspected infected persons within 30 days before screening, or living abroad within 30 days before screening history;
2. Anyone who is allergic to any vaccines, drugs, foods or known excipients (Dlin-MC3-DMA, cholesterol, distearoylphosphatidylcholine, PEG2000-DMG);
3. Have a history of SARS virus infection;
4. Upon questioning, have a history of COVID-19 vaccination, or have received other inactivated vaccines within 14 days before screening, and received live attenuated vaccines within 28 days;
5. Patients have a medical history or family history of epilepsy, convulsions or convulsions, neurological diseases and mental diseases;
6. There are contraindications for intramuscular injection, such as: thrombocytopenia that has been diagnosed, any coagulation disorder or receiving anticoagulant treatment, etc.;
7. The investigator judges that he is known or suspected of having more serious diseases at the same time, including but not limited to: respiratory diseases (tuberculosis, lung failure, etc.), liver and kidney diseases, cardiovascular diseases (heart failure, severe hypertension, etc.), Malignant tumor, infection or allergic skin disease, HIV infection (test report can be provided), or during the active period of acute infection or chronic disease (within 3 days before vaccination);
8. Congenital malformations, developmental disorders, or chronic diseases that the investigator judges are not suitable for participating in this study (such as Downs syndrome, sickle cell anemia or neurological disorders, Guillain-Barre syndrome, etc.), excluding stable diabetes/hypertension );
9. Patients with known immunological impairment or low immunological function diagnosed by the hospital before enrollment, or functional asplenia or splenectomy caused by any situation;
10. There is evidence that they are smokers (smokers >=10 cigarettes/day), alcoholics (alcohol consumption >=4 units/day), drug abusers, and those who do not agree to quit smoking or drinking during the trial;
11. Positive SARS-CoV-2 nucleic acid test and/or positive antibody test before the first dose of vaccine, and/or abnormal imaging examination (small patchy shadow and interstitial change, obvious peripheral lung zone, ground-glass shadow, infiltrating shadow, lung consolidation, etc.), and/or decreased lymphocyte count;
12. Female: those who have a positive blood pregnancy test, are pregnant, breastfeeding, or have a pregnancy plan within one year; men: whose spouse has a pregnancy plan within one year;
13. Patients have participated in other clinical trials (drugs, biological products or devices) within 3 months before the first dose of vaccine, or plan to participate in other clinical trials during the research period;
14. Patients received immune enhancement or immunosuppressive therapy within 6 months before the first dose of vaccine (continuous oral or instillation for more than 14 days);
15. Patients donated blood >=400 ml within 28 days before screening, or received whole blood, plasma and immunoglobulin therapy within 6 months before screening;
16. Currently receiving research drug treatment to prevent COVID-19;
17. Patients are taking antipyretic, analgesic and anti-allergic drugs within 3 days before enrollment;
18. The investigator judges that the subjects cannot follow the research procedures, comply with the agreement, or plan to permanently relocate from the area before the end of the research, or plan to leave the local area for a long time during the scheduled visit period;
19. The relevant staff involved in this study or their immediate family members (such as spouses, parents, siblings or children).
20. According to the investigator's judgment, there are other situations that are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events including solicited adverse event（AE） and unsolicited adverse event（AE） | Solicited AE -14 days post-vaccination, all adverse events other than solicited AE - 28 days after vaccination
  Solicited AE--14 days post-vaccination, common reactions at the vaccination site and non-vaccination site pre-listed on the subject's diary card and electronic case report form（eCRF）, including pain, induration, swelling, rash, flushing, itching, cellulitis at injection site, fever, headache, chills, anorexia, diarrhea, nausea, vomiting, fatigue, weakness, arthralgia, acute allergic reaction, muscle pain at non-inoculation site.
  non-solicited AE --28 days after vaccination, all adverse events other than solicited AE and after 14 days.
Incidence of adverse events associated with the experimental vaccine | 28 days after each dose or full vaccination
  Incidence of adverse events associated with the experimental vaccine within 28 days after each dose or full vaccination.

SECONDARY OUTCOMES:
Incidence of grade ≥3 adverse events | 28 days after each dose or full vaccination
Incidence of grade ≥3 adverse events associated with the experimental vaccine | 28 days after each dose or full vaccination
Withdrawal from the trial due to adverse events | 28 days after each dose or full vaccination
Incidence of serious adverse event（SAE） | 28 days, 3 months, 6 months and 12 months after primary immunization to full immunization
Incidence of SAEs associated with the experiment vaccine | 28 days, 3 months, 6 months and 12 months after primary immunization to full immunization
Incidence of clinically significant abnormalities in laboratory tests | 28 days after each dose or full vaccination

OTHER OUTCOMES:
Positive conversion rate of anti-2019 novel coronavirus S protein-specific antibody (IgG) (average titer increase ≥4 times compared with baseline) | 14 days and 28 days after the first dose；7 days, 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Geometric mean titer (GMT) of anti-2019 novel coronavirus S protein-specific antibody (IgG) and mean fold increase compared with baseline | 14 days and 28 days after the first dose；7 days, 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Positive conversion rate of anti-2019 novel coronavirus neutralizing antibody GMT （average titer increase ≥4 times compared with baseline) | 14 days and 28 days after the first dose；7 days, 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Geometric mean titer (GMT) of anti-2019 novel coronavirus neutralizing antibody and mean fold increase compared with baseline | 14 days and 28 days after the first dose；7 days, 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination
Level of specific cellular immune response against 2019 novel coronavirus（CD4+、CD8+ and IL-2、IL-4、IL-6、IL-10、IFN-γ and TNF-α） | 14 days and 28 days after the first dose, 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after full vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, Principal Investigator — Shulan (Hangzhou) Hospital; Guiling Chen, Principal Investigator — Shulan (Hangzhou) Hospital; Fengli Zhao, Principal Investigator — Yuncheng Central Hospital; Jinlian Bi, Principal Investigator — Xiangya Boai Rehabilitation Hospital
Locations (3):
- China (3):
  - Xiangya Boai Rehabilitation Hospital, Changsha, Hunan
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Chen GL, Yu XY, Luo LP, Zhang F, Dai XH, Li N, Shen ZW, Wu KQ, Lou DF, Peng CG, Jin TH, Huang YM, Shao X, Liu Q, Jiang Q, Guo T, Cao F, Zhu JR, Wu XH, Pei RJ, Deng F, Jiang GP, Li YH, Gao HN, He JX, Zhong-Chen, Peng YC, Li LJ. Phase I study of a non-S2P SARS-CoV-2 mRNA vaccine LVRNA009 in Chinese adults. Vaccine. 2023 Nov 22;41(48):7297-7306. doi: 10.1016/j.vaccine.2023.10.065. Epub 2023 Nov 3. PMID 37925316